CLINICAL TRIAL: NCT06042998
Title: A Prospective, Multicenter, Randomized, Controlled Study of the Clinical Efficacy of Robotic and Laparoscopic Radical Gastrectomy in Neoadjuvant Gastric Cancer Patients
Brief Title: A Multicenter, RCT Study of the Clinical Efficacy of Robotic and Laparoscopic Gastrectomy in Neoadjuvant Gastric Cancer
Acronym: CLASS14
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-14
Record Dates: First submitted 2023-08-02; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Gastric Cancer Stage II; Gastric Cancer Stage III
Keywords: Neoadjuvant therapy; gastric cancer; robot radical gastrectomy; laparoscopic Gastrectomy; short-term clinical outcome; prognosis
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Group A (experimental group): Performing robot radical gastrectomy Group B (control group): Performing laparoscopic radical gastrectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic group (Experimental): Robotic gastrectomy
  Interventions: Procedure: Robotic radical gastrectomy
- Laparoscopic group (Active Comparator): Laparoscopic gastrectomy
  Interventions: Procedure: Robotic radical gastrectomy

INTERVENTIONS:
Procedure: Robotic radical gastrectomy — Laparoscopic gastrectomy
  Other Names: Laparoscopic gastrectomy

SUMMARY:
To evaluate the clinical efficacy of robot radical Gastrectomy and laparoscopic radical Gastrectomy, patients with gastric adenocarcinoma (cT2N+M0 or cT3-4a/N+M0, phase II and III) undergoing neoadjuvant treatment were selected as subjects.

DETAILED DESCRIPTION:
1. Research background In the world, gastric cancer is a common malignant tumor, with the incidence rate ranking fourth and tumor related deaths ranking second. Although the incidence rate of gastric cancer in western countries has a downward trend, it still remains at a high level in East Asia. China is a high incidence area of gastric cancer and a traditional country of gastric cancer. A large number of cases have brought patients a heavy Disease burden.

   Unlike early diagnosis and treatment in developed countries such as Japan and South Korea, gastric cancer in China is mostly diagnosed in the middle to late stage, and the treatment effect is not yet satisfactory. Locally advanced gastric cancer remains the main challenge for the treatment of gastric cancer. The current treatment strategy for locally advanced gastric cancer is a multidisciplinary treatment strategy centered on surgery. Since the MAGIC trial, neoadjuvant chemotherapy for gastric cancer has been widely accepted. Possible advantages of neoadjuvant therapy include better patient tolerance, tumor progression, and elimination of occult micro metastasis to improve radical resection and better prognosis.

   Since the first laparoscopic gastric cancer surgery reported by Kitano et al. in 1994, it has undergone more than 20 years of continuous exploration and innovation. Laparoscopic gastric cancer surgery has rapidly developed worldwide and has now been widely recognized both domestically and internationally. A large number of studies on laparoscopic gastric cancer surgery and laparotomy have confirmed that Laparoscopy has the advantages of less complications, less blood loss during operation, less postoperative pain and inflammatory reaction, rapid recovery of gastrointestinal function, short postoperative hospital stay, and good cosmetic effect, and the oncological treatment effect is equivalent to that of open surgery. At present, laparoscopic surgery for gastric cancer is gradually developing, but the traditional Laparoscopy is limited in fine operation, vision and other aspects. In order to overcome the limitations of laparoscopic surgery, the da Vinci robot system has emerged. As an advanced laparoscopic system, the robot has solved many shortcomings of conventional laparoscopy with its unique advantages. A clearer field of view can better display small anatomical structures, which is conducive to achieving skeletonization of gastric perivascular structures. At the same time, it reduces the difficulty of lymph node dissection and bleeding. At the same time, it has a simulated wrist with 7 degrees of freedom, greatly improving the flexibility of operation and reducing the difficulty of suturing. In the field of gastric cancer surgery, since Hashizume et al. first reported robot gastric cancer surgery in 2002, there have been increasing reports on the safety and feasibility of robot surgical systems applied to gastric cancer treatment. At present, a large number of studies have confirmed that compared with Laparoscopy, robotic surgery can also achieve radical resection, and has the advantages of less intraoperative blood loss and more lymph nodes to be cleared.

   However, the safety and effectiveness of da Vinci surgery are still unclear for patients after neoadjuvant chemotherapy. The pro fibrotic response caused by chemotherapy and the loss of normal tissue planes caused by cytotoxicity pose new technological challenges. Whether less trauma and more lymph node dissection are equivalent to better postoperative safety, chemotherapy completion rate, and survival benefits remains a key issue in clinical practice. Previous RCT studies have shown that LADG seems to provide better postoperative safety and adjuvant chemotherapy tolerance than ODG for locally advanced gastric cancer patients receiving neoadjuvant chemotherapy. Therefore, further targeted research is needed to explore robotic gastric cancer surgery for neoadjuvant therapy.

   Based on the above background, the safety and effectiveness of robotic Gastrectomy in gastric cancer patients undergoing new adjuvant treatment is a key clinical problem in gastric surgery that needs to be solved urgently. Therefore, on the basis of traditional laparoscopy and robotic laparoscopy, this study compared the short-term and long-term clinical efficacy of Leonardo da Vinci Gastrectomy in the neoadjuvant treatment of gastric cancer with gastric adenocarcinoma patients undergoing neoadjuvant treatment.
2. Research Purpose To evaluate the clinical efficacy of robot radical Gastrectomy and laparoscopic radical Gastrectomy, patients with gastric cancer (cT2N+M0 or cT3-4a/N+M0, phase II and III) undergoing neoadjuvant treatment were selected as subjects.
3. Research Design Adopting a multicenter, prospective, open, randomized, controlled, and non-inferiority validation design.

3.2 Comparison and grouping Group A (experimental group): Performing robot radical gastrectomy for gastric cancer Group B (control group): Performing laparoscopic radical gastrectomy for gastric cancer 3.3 Estimation of Sample Size This study used the 3-year disease-free survival rate (DFS) as the main efficacy evaluation indicator. Using 1:1 random grouping, The planned collection of cases is 1.5 years, and the last case will be followed up for another 3 years after enrollment. Due to the lack of previous similar research results, the dual standard method described in Neuenschwander et al.'s paper was used to calculate the required sample size to determine the non disadvantages of robotic versus laparoscopic gastric cancer radical surgery based on DFS [20]. The first criterion is the critical threshold for HR valuation to be less than 1.08, while the second criterion requires that the upper limit of the one-sided 95% confidence interval for non inferiority margin valuation be less than 1.24. The inspection level is taken as 0.05 (bilateral), and the inspection efficiency is taken as 0.8. Using PASS calculation, the sample size N=269, which means that each group requires 268 people. Considering possible exclusion and loss of follow-up cases (10% dropout rate), the final sample size required for each group is 294, with a total of 588 cases required.

3.4 Blind method: This study adopts an open design 3.5 Research cycle Case enrollment cycle: Complete the required case enrollment within 1.5 years. Follow up period: The first case is included as the starting point for follow-up, and the main research purpose is 3 years after the last case is included End point of follow-up. Expected time: June 2023- December 2024 (completion of enrollment) - December 2027 (completion of follow-up) 3.6 Randomization This study adopts a central dynamic randomization method based on minimization, considering stratified factors such as age, BMI, preoperative staging, chemotherapy regimen, and tumor location. After each case is selected, a dedicated person from the participating research center is responsible for inputting the selected case information (age, BMI, preoperative staging, neoadjuvant treatment plan, tumor location) into the central randomization system. The system will immediately return the randomization results to the research center. Researchers from each participating research center should strictly follow the grouping to determine whether the subjects will enter Group A (experimental group) or Group B (control group).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ 75 years old male or female;
2. The primary gastric lesion was diagnosed as gastric adenocarcinoma (papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, Signet ring cell carcinoma, poorly differentiated adenocarcinoma) by endoscopic biopsy histopathology;
3. Before neoadjuvant treatment, the preoperative clinical staging was confirmed to be II and III (cT2N+M0 or cT3-4a/N+M0) through gastroscopy/ultrasound gastroscopy, enhanced CT/MR, or diagnostic laparoscopic exploration (based on AJCC-8th TNM tumor staging);
4. 2-4 cycles of neoadjuvant therapy (chemotherapy+/- targeted/immunotherapy, simple chemotherapy);
5. After new adjuvant treatment, radical Gastrectomy is feasible after MDT discussion;
6. Preoperative ECOG physical condition score of 0/1 or Karst score ≥ 70%;
7. Preoperative ASA score I-III;
8. The expected survival period exceeds 6 months;
9. Willing and able to comply with the research protocol;
10. Sign a written informed consent form before enrollment and be fully aware of the right to withdraw from this study at any time.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Suffering from serious mental illness;
3. History of upper abdominal surgery (excluding history of laparoscopic cholecystectomy);
4. History of gastric surgery (excluding ESD/EMR for gastric cancer);
5. Moderate to severe renal insufficiency;
6. Organ transplant recipients receiving immunosuppressive therapy;
7. Have a history of other malignant diseases within 5 years;
8. Have a history of unstable angina or myocardial infarction within 6 months;
9. Have a history of cerebral infarction or cerebral hemorrhage within 6 months;
10. Have a history of continuous systemic corticosteroid therapy within one month;
11. Simultaneous surgical treatment of other diseases is required (excluding laparoscopic cholecystectomy);
12. Gastric cancer comorbidities (bleeding, perforation, obstruction) requiring emergency surgery;
13. Lung function test FEV1<50% of expected value;
14. The patient has participated or is currently participating in other clinical studies (within 6 months).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | three years after surgery
  3-year disease-free survival

SECONDARY OUTCOMES:
3-year overall survival rate | three years after surgery
  3-year overall survival rate
overall postoperative morbidity rates | 30 days after surgery
  overall postoperative morbidity rates
postoperative recovery course | 14 days surgery
  postoperative recovery course

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastrointestinal Surgery, Qingdao University Affiliated Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided
Sharing data with participating centers